CLINICAL TRIAL: NCT06540885
Title: A Comparison Between Palonosetron Versus Granisetron As Postoperative Nausea and Vomiting Prophylaxis In Idiopathic Scoliosis Surgery: A Randomized Control Trial
Brief Title: A Comparison Between Palonosetron Versus Granisetron as PONV Prophylaxis in Scoliotic Patients Undergoing Spine Surgery
Acronym: PONV
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Siti Nadzrah Yunus, Doctor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202464-13794
Record Dates: First submitted 2024-06-10; First posted 2024-08-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Nausea and Vomiting; Scoliosis
Keywords: Antiemetics; Granisetron; Palonosetron
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Scoliosis | interventions — Palonosetron; Antiemetics; Granisetron

STUDY DESIGN:
Intervention Model Description: After taking informed consent and recruitment of eligible participants, they will be randomized using a sequentially numbered, opaque sealed envelope (SNOSE) method. 74 radio-opaque envelopes will be prepared according to two groups: 37 participants for each Palonosetron Group (Group P) and Granisetron Group (Group G). Group P will receive Intravenous (IV) palonosetron 1.5mcg/kg prior to the commencement of general anaesthesia; while Group G) will receive IV granisetron 1mg at the start of wound closure.
Who Masked: Participant, Investigator
Masking Description: All the anaesthesiologists and patients involved in the study were blinded to group allotment. Patient allotment will be revealed prior to the surgery via the sealed envelope to an anaesthetic nurse or doctor (who is not involved in study) for drug preparation. Participants will receive 2 separate injections of the study drugs/placebo. The first injection given prior to commencement of general anaesthesia comprises of palonosetron 1.5mcg/kg (maximum dose of 75mcg) diluted with normal saline 0.9% to make up a 5ml preparation (for Group P), or a 5ml preparation of normal saline 0.9% as placebo (for Group G). The second injection will be administered at the start of wound closure, comprising either 5ml of preparation of normal saline 0.9% as placebo (for Group P), or IV Granisetron 1mg diluted into a 5ml preparation of normal saline 0.9% for Group G.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palonosetron Group (Group P) (Experimental): Group P will receive a stat dose of IV palonosetron 1.5mcg/kg diluted in a 5ml preparation of normal saline 0.9% prior to the commencement of general anaesthesia. At the start of wound closure, Group P will receive a 5ml preparation of normal saline 0.9% as a placebo.
  Interventions: Drug: Palonosetron (Group P)
- Granisetron Group (Group G) (Active Comparator): Group G will receive a 5ml preparation of normal saline 0.9% as placebo prior to commencement of general anaesthesia. At the start of wound closure, a stat dose of IV granisetron 1mg in 5ml preparation will be administered.
  Interventions: Drug: Granisetron (Group G)

INTERVENTIONS:
Drug: Palonosetron (Group P) — Group P will be receiving palonosetron 1.5mcg/kg before the commencement of general anaesthesia
  Other Names: antiemetic
  Arms: Palonosetron Group (Group P)
Drug: Granisetron (Group G) — Group G participants will receive IV Granisetron 1mg at the start of wound closure
  Other Names: antiemetic
  Arms: Granisetron Group (Group G)

SUMMARY:
The aim of this clinical trial is to compare the effectiveness of two Serotonin (5- HT3) receptor antagonist, palonosetron and granisetron, administered along with dexamethasone as a preventive measure against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent patients with idiopathic scoliosis (IS) undergoing posterior spinal fusion (PSF) surgery under total intravenous anesthesia (TIVA).

The main questions the study aims to answer are:

How effective is palonosetron compared to granisetron, when both combined with dexamethasone, in preventing PONV after scoliosis surgery? Are there any differences in the need for rescue antiemetics, occurrence of adverse effects related to the study drugs, and patient satisfaction between the two treatment groups? Participants in the study will be randomly assigned to receive either palonosetron or granisetron in addition to dexamethasone as part of their anesthesia and antiemetic regimen. The incidence and/ or severity of nausea, vomiting and retching will be assessed at 1 hour, 4 hours, 12 hours, 24 hours and 48 hours after surgery.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) remains a common adverse event after surgery and anaesthesia causing much dissatisfaction among patients. PONV incidence is reported at 30% in all surgical patients and up to 80% in high-risk patients. Idiopathic scoliosis is a common form of structural spinal deformities with a Cobb angle of >/ 10 degrees. It affects young females in the early pubertal stage more than young men by 1% and 4%.

Posterior spinal fusion (PSF) surgery is commonly performed in patients with severe scoliosis. It is a long complex surgery inflicting extensive surgical field requiring opioids as the mainstay of analgesia during the perioperative period. These targeted population are particularly adolescent female requiring intraoperative and postoperative opioids who are at high risk of developing PONV.

Dexamethasone and anti-serotonergic drugs like granisetron are commonly used antiemetics due to their efficacy and safety profiles. Dexamethasone is particularly favoured for its long duration of action and pain-reducing effects.

Palonosetron, a second-generation anti-serotonergic drug, has a unique pharmacokinetic profile with a prolonged duration of action. It may be more beneficial for patients on prolonged opioid-based analgesic regimens. However, its higher cost and inconsistent study findings limit its widespread use, especially in scoliosis patients undergoing spinal fusion surgery.

Total intravenous anaesthesia (TIVA) is recommended for high-risk PONV patients, as it reduces the emetogenic effect of volatile anaesthetics. Propofol, used in TIVA, is itself an effective antiemetic. TIVA with propofol has been shown to be as effective as giving a single antiemetic and can further reduce the risk of PONV when combined with other prophylactic antiemetics.

The standard practice for managing PONV involves the administration of two antiemetics and considering TIVA for high-risk patients. This study aims to compare the effectiveness of palonosetron and ondansetron when administered alongside dexamethasone in scoliosis patients undergoing spinal fusion under TIVA. The study will also evaluate the number of rescue antiemetics needed, assess adverse effects, and measure patient satisfaction.

The study will be randomized and double-blinded, to be conducted in University Malaya Medical Centre (UMMC). The sample size is calculated to be 92 participants, after taking into account a 20% dropout rate. Adult and adolescent idiopathic scoliosis patients undergoing PSF surgery will be eligible for the study. Written informed consent will be obtained from participants or their guardians, and assent will be obtained from adolescent participants. Patients will be randomized to receive either palonosetron or ondansetron along with dexamethasone.

The study will follow standard anaesthetic techniques, including TIVA with remifentanil and propofol. Intravenous injections of the study drugs or placebo will be given during surgery, and dexamethasone will be administered as a baseline antiemetic. Morphine will be administered before the end of surgery for pain management.

ELIGIBILITY:
Inclusion Criteria:

* Age: 10 years and above
* American Society of Anesthesiologists (ASA) class I-II

Exclusion Criteria:

* Active smoker
* Obesity with body mass index (BMI) of 34 and above
* Body weight of less than 30kg
* History of gastro-esophageal reflux disease (GERD)/ other gastrointestinal diseases associated with vomiting
* History of motion sickness
* History of allergy to 5-HT3 (serotonin) receptor antagonists or dexamethasone
* History of nausea or vomiting withing 24 hours before surgery
* History of administration of antiemetics/ steroids/ psychoactive medications within 24 hours before the surgery
* History of cardiac arrhythmias
* Prolonged QT (QTc is prolonged if > 430ms in men or >450ms in women)

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV) delayed postoperative nausea and vomiting (PONV) in adult and adolescent idiopathic scoliosis patients | At 1 hour after surgery
  To compare the effectiveness of palonosetron and granisetron when administered alongside dexamethasone as prophylaxis against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent idiopathic scoliosis patients undergoing posterior spinal fusion surgery under total intravenous anaesthesia.
Incidence of postoperative nausea and vomiting (PONV) | At 4 hours after surgery
  To compare the effectiveness of palonosetron and granisetron when administered alongside dexamethasone as prophylaxis against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent idiopathic scoliosis patients undergoing posterior spinal fusion surgery under total intravenous anaesthesia.
Incidence of postoperative nausea and vomiting (PONV) | At 12 hours after surgery
  To compare the effectiveness of palonosetron and granisetron when administered alongside dexamethasone as prophylaxis against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent idiopathic scoliosis patients undergoing posterior spinal fusion surgery under total intravenous anaesthesia.
Incidence of postoperative nausea and vomiting (PONV) | At 24 hours after surgery
  To compare the effectiveness of palonosetron and granisetron when administered alongside dexamethasone as prophylaxis against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent idiopathic scoliosis patients undergoing posterior spinal fusion surgery under total intravenous anaesthesia.
Incidence of postoperative nausea and vomiting (PONV) | At 48 hours after surgery
  To compare the effectiveness of palonosetron and granisetron when administered alongside dexamethasone as prophylaxis against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent idiopathic scoliosis patients undergoing posterior spinal fusion surgery under total intravenous anaesthesia.

SECONDARY OUTCOMES:
To evaluate the need for rescue antiemetics among participants | At 1 hour, 4 hours, 12 hours, 24 hours and 48 hours after surgery
  Number of Participants Developing Postoperative Nausea Vomiting Requiring Rescue Antiemetic Within 48 hours After Surgery Any occurrence of severe nausea and retching with visual analogue scale score ≥4; and vomiting of 1 or more episodes will be treated with the rescue drug IV metoclopramide. For adolescent subjects (aged less than 18 years old), IV metoclopramide will be given at 0.2mg/kg, with a maximum dose of 10 mg intravenously up to 3 times per day. For adult patients (18 years old and above), IV metoclopramide 10mg will be given, up to 3 times per day. If there is any further occurrence of PONV within 8 hours of administration of IV metoclopramide, a second line of rescue antiemetic, IV Granisetron 1mg, will be administered to participants in both arms of the study. The administration of any rescue medications will be recorded and taken into account during data processing.
To evaluate the adverse effects related to the study drugs. | At 1 hour, 4 hours, 12 hours, 24 hours and 48 hours after surgery
  Number of Participants Developing Adverse Effects Related to the Study Drugs.
To assess the degree of participant's satisfaction. | At 48 hours after surgery
  Degree of patient satisfaction as represented on the Likert scale Selection of a number from a scale of 1 (least satisfied) to 5 (most satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Nantni Kumaran, MBBS, Principal Investigator — University of Malaya; Mohd Shahnaz Hasan, MAnaes, MBBS, Principal Investigator — University of Malaya
Locations (2):
- Malaysia (2):
  - University Malaya, Pantai Valley, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cao X, White PF, Ma H. An update on the management of postoperative nausea and vomiting. J Anesth. 2017 Aug;31(4):617-626. doi: 10.1007/s00540-017-2363-x. Epub 2017 Apr 28. PMID 28455599
- [Result] Johansson E, Hultin M, Myrberg T, Wallden J. Early post-operative nausea and vomiting: A retrospective observational study of 2030 patients. Acta Anaesthesiol Scand. 2021 Oct;65(9):1229-1239. doi: 10.1111/aas.13936. Epub 2021 Jul 4. PMID 34086350
- [Result] Cheng JC, Castelein RM, Chu WC, Danielsson AJ, Dobbs MB, Grivas TB, Gurnett CA, Luk KD, Moreau A, Newton PO, Stokes IA, Weinstein SL, Burwell RG. Adolescent idiopathic scoliosis. Nat Rev Dis Primers. 2015 Sep 24;1:15030. doi: 10.1038/nrdp.2015.30. PMID 27188385
- [Result] Schraag S, Pradelli L, Alsaleh AJO, Bellone M, Ghetti G, Chung TL, Westphal M, Rehberg S. Propofol vs. inhalational agents to maintain general anaesthesia in ambulatory and in-patient surgery: a systematic review and meta-analysis. BMC Anesthesiol. 2018 Nov 8;18(1):162. doi: 10.1186/s12871-018-0632-3. PMID 30409186
- [Result] Schaefer MS, Kranke P, Weibel S, Kreysing R, Kienbaum P. Total intravenous anaesthesia versus single-drug pharmacological antiemetic prophylaxis in adults: A systematic review and meta-analysis. Eur J Anaesthesiol. 2016 Oct;33(10):750-60. doi: 10.1097/EJA.0000000000000520. PMID 27454663
- [Result] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Result] Marret E, Kurdi O, Zufferey P, Bonnet F. Effects of nonsteroidal antiinflammatory drugs on patient-controlled analgesia morphine side effects: meta-analysis of randomized controlled trials. Anesthesiology. 2005 Jun;102(6):1249-60. doi: 10.1097/00000542-200506000-00027. PMID 15915040
- [Result] Elia N, Lysakowski C, Tramer MR. Does multimodal analgesia with acetaminophen, nonsteroidal antiinflammatory drugs, or selective cyclooxygenase-2 inhibitors and patient-controlled analgesia morphine offer advantages over morphine alone? Meta-analyses of randomized trials. Anesthesiology. 2005 Dec;103(6):1296-304. doi: 10.1097/00000542-200512000-00025. PMID 16306743